CLINICAL TRIAL: NCT06012682
Title: A Randomized, Controlled, Double-blind Study Clinical Trials Evaluating the Effect of Metformin Treatment on Function Endometrium in Women Diagnosed With Idiopathic Infertility
Brief Title: Clinical Trials Evaluating the Effect of Metformin Treatment on Function Endometrium in Women Diagnosed With Idiopathic Infertility
Acronym: METIN
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021/ABM/03/00006
Record Dates: First submitted 2023-06-22; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- metformin (Experimental): patients randomized to received metformin
  Interventions: Drug: Metformin Hydrochloride
- placebo (Placebo Comparator): patients randomized to received placebo
  Interventions: Drug: Placebo
- group without intervention (No Intervention)

INTERVENTIONS:
Drug: Metformin Hydrochloride — The investigational medicinal product/placebo will be dispensed to study participants by study staff during randomization visits V1, V2, V3, V4, V5 and V6.
  The randomized patient will receive the investigational medicinal product/placebo in tablets of 500 mg. The received tablets will be dispensed in an amount sufficient for the next visit. Patients will be asked to bring unused medicine and all empty ones packaging to the Center for each subsequent visit. The investigational medicinal product/placebo will be administered orally 500 mg three times a day (Table No. 1). The dose of the study product will be gradually increased from 500 mg/day to 1500 mg/day in order to avoid or reduce side effects related to taking the study medicinal product metformin
  Arms: metformin
Drug: Placebo — The investigational medicinal product/placebo will be dispensed to study participants by study staff during randomization visits V1, V2, V3, V4, V5 and V6.
  The randomized patient will receive the investigational medicinal product/placebo in tablets of 500 mg. The received tablets will be dispensed in an amount sufficient for the next visit. Patients will be asked to bring unused medicine and all empty ones packaging to the Center for each subsequent visit. The investigational medicinal product/placebo will be administered orally 500 mg three times a day (Table No. 1). The dose of the study product will be gradually increased from 500 mg/day to 1500 mg/day in order to avoid or reduce side effects related to taking the study medicinal product metformin
  Arms: placebo

SUMMARY:
Randomized, controlled, double-blind, three-arm clinical trial in which 75 women will be randomized to treatment with metformin, 75 women to treatment with placebo and 50 women to the observation group. The medical intervention will last 24 weeks (6 months). Women with confirmed idiopathic infertility, in whom infertility factors have been excluded during full diagnostics, will be included in the study

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45
2. No pregnancy for a minimum of 12 months prior to screening.
3. Diagnosed with idiopathic infertility.
4. No use of hormone therapy 30 days before screening.
5. No use of any methods of contraception 30 days before screening and during the examination.
6. BMI between 18.5 - 30 kg/m2.

Exclusion Criteria:

1. Positive pregnancy test result.
2. Patients diagnosed with another factor of infertility.
3. Patients with type I or II diabetes.
4. Patients taking metformin or other hypoglycaemic drugs in the last 4 weeks before screening.
5. Patients with hepatic impairment and abnormal liver function tests (alanine aminotransferase and/or aspartate aminotransferase (above 3x ULN).
6. Patients with an eGFR less than 45 mL/min/1.73m2.
7. Accompanying chronic diseases with poor prognosis.
8. Patients with a history of lactic acidosis or other metabolic acidosis.
9. Patients with a history of congestive heart failure III/IV NYHA degree.
10. Patients with acute myocardial ischemia.
11. Patients with sepsis or severe infection.
12. Diseases which, in the opinion of the investigator, constitute an exclusion criterion and prevent the patient from participating in the study.
13. Patients with predictable problems with cooperation with the research team.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Effects of metformin on fertility and the possibility of becoming pregnant,as measured by pregnancy test strips and β-hCG levels | 4 years
  The aim of the study is to evaluate the effect of metformin on endometrial function in women diagnosed with idiopathic infertility, by proving the use of the proposed therapy to improve fertility in these women.

SECONDARY OUTCOMES:
Evaluation of the effect of metformin therapy on endometrial function. | 4 years
  It will be tested by assessing the concentration of biomarkers in the tissue before and after treatment
Molecular analysis of endometrial tissues using Next Generation Sequencing (NGS) technology | 4 years
  Transcriptome analysis of endometrial tissues before and after metformin therapy.
Intra-tissue metabolic profiling of steroids | 4 years
  The study will test whether treatment with metformin affects the intracrine production of steroid hormones in the endometrium.
Oxidative stress evaluation by using total oxidative capacity (TOC) and total antioxidant capacity (TAC) | 4 years
  In-depth analysis of molecular and cellular processes using multi-omics combined with clinical data will provide essential knowledge about the mechanisms of metformin's action, which may have clinical applications not only in cases of idiopathic female infertility but also in other disorders.
Quality of Life questionary evaluation SF-36, FertiQoL, | 24 weeks
  The results on the response scales are rotatable, summed and scaled from 0 to 100. Subscale and higher scores indicate good quality life. The number of obtained equation points is 50 or less arrangements with a psychologist.